CLINICAL TRIAL: NCT01059162
Title: Evaluation of OT-135P (IOPtiMateTM) : Beam Manipulating System for CO2 Laser Assisted Non-Penetrating Glaucoma Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IOPtima Ltd. (Industry)
Responsible Party: Dan Peres, COO, IOPtima Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCL-34-003 (03)
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Open Angle Glaucoma; Pseudo-Exfoliative Glaucoma
Keywords: Glaucoma Surgery; Filtering Surgery; Non Penetrating glaucoma surgery
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IOPtiMate (Experimental): patients will undergo non-penetrating laser assisted filtering surgery by the IOPtiMate (OT-134) system
  Interventions: Device: Laser Assisted Non-penetrating glaucoma surgery

INTERVENTIONS:
Device: Laser Assisted Non-penetrating glaucoma surgery — A layer by Layer ablation of the deep sclera (under the superficial scleral flap) to achieve functional fluid percolation of the inner eye humor without penetration.

SUMMARY:
The aim of the study is to evaluate the safety and effectiveness of the IOPtiMate (OT-135P) in Laser Assisted Non-Penetrating Glaucoma surgery in Open-Angle and Pseudoexfoliative Glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be 18 years of age or older.
2. Patient must have primary open angle glaucoma or pseudo-exfoliative glaucoma in the study eye; diagnosis is based on glaucomatous optic neuropathy, Shaffer angle of +2 and visual field defect attributed to glaucoma (at least two consecutive abnormal visual field test results, defined as a pattern SD (PSD) outside the 95% normal confidence limits and/or glaucoma Hemifield Test (Carl Zeiss Meditec, Inc.).
3. Eye to be treated must be phakic or pseudophakic eye with no ocular disorder or ocular diseases but cataract, and no prior surgical intervention in study eye but cataract surgery with clear corneal incision and trabeculoplasty performed > 3 months ago.
4. Patient is indicated for filtration surgery.
5. Presence of ocular hypertension, defined as an intraocular corrected pressure (IOP) ≥ 21 mm Hg in the study eye, while on maximal tolerated medications . This IOP level of above or equal 21 mmHg must be verified and recorded in the most recent 2 consecutive measurements (but not taken on the same day) prior to operation.
6. Best corrected visual acuity (BCVA) better than 20/200 in the fellow eye.
7. Optic neuropathy is attributed exclusively to glaucoma.
8. Patient or legal guardian agrees to sign written informed consent prior to study participation.
9. Patient is able and willing to complete post-operative follow-up requirements.

Exclusion Criteria:

1. Patient has previously undergone a non-penetrating glaucoma surgery with the IOPtima CO2 Laser System in fellow eye.
2. Diagnosis of glaucoma other than primary open angle glaucoma or pseudo-exfoliative glaucoma.
3. History of previous intraocular surgery in the study eye; referring to but not limited to glaucoma filtering surgery (penetrating and non-penetrating), laser gonioplasty, corneal transplant, and history of any other laser ocular procedures except for laser trabeculoplasty surgery.
4. Laser trabeculoplasty surgery within the last three months in the study eye.
5. Study eye is aphakic.
6. Patients with previous cataract extraction with scleral tunnel and or conjunctival incision in the study eye.
7. Proliferative or severe non-proliferative retinopathy in either eye.
8. Eyes with (dilated) pupil diameter of less than 2 mm in the study eye.
9. Discernable congenital anomaly of the anterior chamber angle in the study eye.
10. Patients with neuropathy other than glaucoma in the study eye.
11. Patient with RVO (retinal vein occlusion) in the study eye.
12. Patient with RAO (retinal artery occlusion) in the study eye.
13. History of prior vitrectomy or Vitreous Hemorrhage (VH) in the study eye.
14. Patient with media opacification which may interfere with optic nerve evaluation in the study eye.
15. Patient with a history of severe eye trauma in the study eye
16. Patient with ocular malformations such as microphthalmia in the study eye.
17. Patient with concurrent inflammatory / infective eye disorder (e.g. episcleritis, scleritis) in the study eye
18. Patient with any sign of past or present uveitis (anterior / posterior)
19. Patient with known allergy to the study medications.
20. Patient with severe systemic disease or disabling conditions such as: chronic renal failure requiring dialysis, severe and disenabling neurological disease, and post organ transplants.
21. Patient participating in another clinical trial or participation in another clinical trial is < 3 months.
22. Patient is pregnant or breast feeding. Women of child bearing age will submit a urine sample result for β-HCG (Pregnancy test) within 2 weeks of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Intra-Ocular Pressure (IOP) | 6 months

SECONDARY OUTCOMES:
Number of anti-Glaucoma Medications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Noa Geffen, Dr., Principal Investigator — Glaucoma service, Ophthalmology ward, Meir Hospital, Kfar-Saba; Shlomo Melamed, Dr., Principal Investigator — Glaucoma service, Ophthalmology ward, Sheba Hospital, Tel-Hashomer Israel
Locations (1):
- Ophthalmology ward, Meir Hospital, Kfar Saba, Israel